CLINICAL TRIAL: NCT00612079
Title: The Effect of Sertindole on Sensory Gating and Cognition in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other); H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 97_PPI-P50; E-07/2007; 2007DR1251
Record Dates: First submitted 2008-01-23; First posted 2008-02-11 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Sertindole; sensory gating; PPI; P50 suppression; CANTAB; Effect of Sertindole on sensory gating (P50 suppression); on sensorimotor gating (PPI); and cognition (CANTAB)
MeSH Terms: interventions — sertindole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Healthy volunteers with high sensory gating levels.
  Interventions: Drug: Sertindole; Drug: Placebo
- 1 (Experimental): Healthy volunteers with low sensory gating levels.
  Interventions: Drug: Sertindole; Drug: Placebo

INTERVENTIONS:
Drug: Sertindole — oral 3 x 4mg
Drug: Placebo — 3 x 4mg Placebo

SUMMARY:
This study aims to further validate and extend our previous findings insofar that the effect of the atypical antipsychotic and mixed 5-HT2/D2 antagonist sertindole on sensorimotor gating processes and its relationship to cognitive performance shall be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Gender: male

Exclusion Criteria:

* Axis I Disorders: lifetime DSM IV diagnosis according to DIA-X of alcohol or illicit drug dependence. No life-time DSM IV diagnosis according to DIA-X of a major affective, psychotic, anxiety disorder, eating-disorder as defined above.
* Axis II Disorders: lifetime DSM IV diagnosis of personality disorder according to SCID-II.
* Family history: lifetime history of 1st degree relative (parents and siblings) of a major affective, psychotic, or anxiety disorder as defined above.
* ECG: QTc-interval >450 msec.
* Systolic blood pressure <100 mmHg
* Bradycardia (Hf < 50/Min) und Arrhythmias
* Hypokalemia or Hypomagnesemia

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Sensory (EEG: P50 suppression) and sensorimotor gating (EMG: PPI) | after placebo and and after medical treatment

SECONDARY OUTCOMES:
Cognitive performances | after placebo and and after medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Franz X. Vollenweider, Prof. Dr. med., Principal Investigator — University Hospital of Psychiatry, Department Neuropsychopharmacology and Brain Imaging
Locations (1):
- University of Psychiatry Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Holstein DH, Csomor PA, Geyer MA, Huber T, Brugger N, Studerus E, Vollenweider FX. The effects of sertindole on sensory gating, sensorimotor gating, and cognition in healthy volunteers. J Psychopharmacol. 2011 Dec;25(12):1600-13. doi: 10.1177/0269881111415734. Epub 2011 Sep 2. PMID 21890590